CLINICAL TRIAL: NCT01439919
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Assess the Clinical Benefit of SSR411298 as Adjunctive Treatment for Persistent Cancer Pain
Brief Title: A Clinical Trial to Assess the Clinical Benefit of SSR411298 as Adjunctive Treatment for Persistent Cancer Pain
Acronym: ACT11705
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to strategic reasons
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT11705; 2011-002557-56 (EudraCT Number); U1111-1115-3390 (Other: UTN)
Record Dates: First submitted 2011-09-07; First posted 2011-09-23 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Pain; Breakthrough Cancer Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SSR411298 200 mg (Experimental): SSR411298 200 mg, one tablet once daily for 4 weeks
  Interventions: Drug: SSR411298
- Placebo (Placebo Comparator): Placebo (for SSR411298), one tablet once daily for 4 weeks
  Interventions: Drug: Placebo (for SSR411298)

INTERVENTIONS:
Drug: SSR411298 — Form: tablet
  Route: oral administration with food
  Arms: SSR411298 200 mg
Drug: Placebo (for SSR411298) — Form: tablet
  Route: oral administration with food
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of SSR411298 200 mg daily compared to placebo as adjunctive treatment for persistent cancer pain based on Numeric Rating Scale (NRS).

Secondary Objectives are:

* To evaluate the effect of SSR411298 200 mg daily on pain, breakthrough pain frequency, background therapy utilization, mood, patient satisfaction of pain relief, nausea, constipation, healthcare utilization and quality of life;
* To evaluate the tolerability and safety of SSR411298 as adjunctive treatment for persistent cancer pain;
* To characterize patient disease, in terms of cancer, cancer treatment, cancer pain and cancer pain treatment;
* To evaluate the pharmacokinetic (PK) exposure of SSR411298 as adjunctive treatment for persistent cancer pain;
* To assess endocannabinoid plasma concentrations.

DETAILED DESCRIPTION:
The total study duration for a participant is 6 weeks (1-week screening, 4-week treatment and 1-week post-treatment follow-up).

Participants continue to receive WHO Step 2 or 3 cancer pain treatment as background therapy.

ELIGIBILITY:
Inclusion criteria:

Patient with moderate or severe, persistent cancer pain who is receiving the World Health Organization (WHO) Step 2 or 3 cancer pain treatment:

* Pain generator (source of pain) must be primarily due to underlying cancer or cancer treatment;
* Pain generator (source of pain) must be classified as either primarily nociceptive or primarily neuropathic;
* Pain severity must be moderate or severe with an average NRS score ≥4 during the screening week.

Exclusion criteria:

* Instability of pain during the screening week;
* Use of prohibited adjuvant pain treatment in the week prior to study entry or plan to use these medications during the study;
* Current use of medication containing tetrahydrocannabinol (THC);
* Chemotherapy within 4 weeks before study entry or chemotherapy planned during the study (a stable regiment of hormonal therapy is permitted);
* Radiotherapy within 4 weeks before study entry or radiotherapy planned during the study (hemostatic palliative radiotherapy is permitted);
* Cancer related surgery within 4 weeks before study entry or cancer-related surgery planned during the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average Numeric Rating Scale (NRS) pain intensity score | 5 weeks (from D-7 (seven days before randomization) up to D28)
  The NRS is an 11-category descriptive anchor scale that is one of the most frequently employed and accepted scales for pain evaluation. Score ranges from 0 [no pain] to 10 [worst possible pain].
  Average NRS score is defined as the average of pain intensity scores measured daily by NRS during a week.

SECONDARY OUTCOMES:
Change from baseline in Brief Pain Inventory Short-Form (BPI-SF) scores | 5 weeks (from D-7 (seven days before randomization) up to D28)
  The BPI-SF is a 9-point questionnaire that measures the intensity of pain, interference of pain, pain relief, pain quality, and patient perception of the cause of pain.
Responder rates | 5 weeks (from D-7 (seven days before randomization) up to D28)
  Responders are defined as:
  * reduction from baseline ≥30% of pain intensity as measured by NRS;
  * reduction from baseline ≥50% of pain intensity as measured by NRS;
  * composite of decrease in pain intensity or decrease in background therapy utilization.
Breakthrough pain frequency | 5 weeks (from D-7 (seven days before randomization) up to D28)
Opioid consumption expressed as the morphine-equivalent dose per day | 5 weeks (from D-7 (seven days before randomization) up to D28)
Rescue medication consumption expressed as the number of rescue medication doses per day | 5 weeks (from D-7 (seven days before randomization) up to D28)
Mood disorders as measured by the Hospital, Anxiety & Depression Scale (HADS) | 5 weeks (from D-7 (seven days before randomization) up to D28)
  The HADS is a self-reported scale that contains 14 items rated on 4-point Likert scales. Two subscales assess depression (7 items) and anxiety (7 items). Each 7-item subscale yields a score of 0 to 21 that is interpreted with the following cut points: 0-7, normal; 8-10, mild mood disturbance; 11-14, moderate mood disturbance; and 12-21, severe mood disturbance.
Change in nausea as measured by Visual Analog Scale (VAS) | 5 weeks (from D-7 (seven days before randomization) up to D28)
  The nausea VAS is a patient-centered instrument to measure nausea on a continuous 100-mm scale.
Constipation as measured by the Bowel Function Index (BFI) | 5 weeks (from D-7 (seven days before randomization) up to D28)
  The BFI is a 3-item questionnaire to measure constipation from the patient's perspective. The time frame for the questions is "during the last 7 days". The answer for each of the 3 items is rated on a scale from 0 (easy or no difficulty) to 100 (severe difficulty).
Healthcare utilization | 5 weeks (from D-7 (seven days before randomization) up to D28)
  Healthcare utilization is measured as the number unscheduled hospitalizations, emergency department visits, healthcare provider office visits, and sick leave days.
Patient satisfaction of pain relief | 5 weeks (from D-7 (seven days before randomization) up to D28)
  Patient satisfaction of pain relief is a 5-point Likert scale that measures patient satisfaction with treatment. The five categorical responses are: extremely unsatisfied, unsatisfied, neutral, satisfied, extremely satisfied.
Quality of life as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) version 3 | 5 weeks (from D-7 (seven days before randomization) up to D28)
  The EORTC QLQ-C30 questionnaire contains a total of 30 items, of which 28 items are rated on 4-point Likert-type scale and 2 items are rated on 7-point Likert scale. These include 5 functional scales, 3 symptom scales, a global health status/QoL scale, and 6 single items.
  A high scale score represents a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Overview of adverse events (AE) | up to 5 weeks (from 1st study drug intake up to 7 days after last study drug intake)
SSR411298 plasma concentration | predose and 3-5 hours after study drug intake on Day D14 and Day 28
  Plasma concentrations of SSR411298 will be determined by a validated liquid chromatography method coupled with tandem mass spectrometry (LC-MS/MS) with a lower limit of quantification (LLOQ) of 10 ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- United States (2):
  - Investigational Site Number 840006, Flat Rock, North Carolina
  - Investigational Site Number 840005, Canton, Ohio